CLINICAL TRIAL: NCT01264224
Title: A Dose-block Randomized, Double-blind, Placebo-controlled Single/Multiple Dosing, Dose-escalation Phase I Clinical Trial to Investigate the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of PAC-14028 After Oral Administration in Healthy Male Volunteers.
Brief Title: PAC-14028 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: AP-TRPV1-PI-01
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — N-(1-(3,5-difluoro-4-methanesulfonylaminophenyl)ethyl)-3-(2-propyl-6-trifluoromethylpyridine-3-yl)acrylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- PAC-14028 (Experimental)
  Interventions: Drug: PAC-14028

INTERVENTIONS:
Drug: PAC-14028 — tablets, oral administration, single/multiple dosing, dose escalation

SUMMARY:
1. Primary Objective:

   * To evaluate safety and tolerability of single and multiple oral dosing of PAC-14028 in healthy male volunteers.
2. Secondary Objective:

   * To evaluate pharmacokinetics and pharmacodynamics of single and multiple oral dosing of PAC-14028 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men aged 20 to 45 years at the time of screening
2. Whose weight is 50kg or more, but less than 90 kg, and whose body mass index(BMI) is 19.0 kg/m^2 or more but less than 27 kg/m^2

   -BMI (kg/m^2) = weight(kg) /{height(m)}^2
3. Who voluntarily decides study participation after receiving detailed explanation about the study and fully understanding it and who provides written consent for compliance with study requirement including proper contraception.

Exclusion Criteria:

1. Who has clinically significant medical history or diseases involving liver, kidney, neurological system, respiratory system, endocrine system, urinary system, cardiovascular system, psychical disorders or blood tumor
2. Who has gastrointestinal diseases or operation history which may interfere study drug absorption (however, except simple appendectomy and hernioplasty )
3. Who has a history of hypersensitivity or allergies to any drug (aspirin, antibiotics, etc)
4. Who has taken any prescribed drugs, herbal agents or crude drugs within 2 weeks before study drug administration, or who has taken any over-the-counter (OTC) drugs or vitamins (Investigators will determine his eligibility by considering the effect of the drug on his safety or pharmacokinetic results in case other inclusion/exclusion criteria is satisfied.)
5. Who has drug abuse history or positive result at urine screening tests (cannabinoid, opioid, amphetamine, cocaine, barbiturate, benzodiazepine)
6. Smoker or who has stopped smoking within previous 1 month or shows positive result at cotinine test.
7. Who has confirmed positive at serological tests (HBs antigen, HCV antibody and HIV antibody)
8. Who consistently consumes alcohol (over 21 units/week, 1 unit = 10 g of pure alcohol)
9. Who has participated in other clinical study within 12 weeks before study drug administration (however, the last dosing day is considered as the end of clinical study.)
10. Who has had bleeding or blood collection and donation over 400 mL within 12 weeks before study drug administration
11. Whose vital sign measured at sitting position after resting at least 5 minutes is as following

    * Low blood pressure (Systolic pressure: 90 mmHg or less, Diastolic pressure: 50 mmHg or less)
    * High blood pressure (Systolic pressure: 140 mmHg or higher, Diastolic pressure: 90 mmHg or less)
12. Who is determined ineligible for study participation by investigators for any reason including clinical lab test and ECG results.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability
  AE incidence pattern, abnormal findings in vital sign, ECG test, and clinical lab tests

SECONDARY OUTCOMES:
Pharmacokinetics/dynamics
  * PK:Concentration of PAC-14028 in Blood and Urine; Cmax, AUC
  * PD:Heat pain threshold/tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University Hospital, Clinical Trials Center/Clinical Research Institute
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea